CLINICAL TRIAL: NCT01244295
Title: Complicated Grief Treatment in Older Adults
Brief Title: Study of Interpersonal Therapy and Complicated Grief Treatment in Adults 50 Years and Older
Acronym: CGTOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5645; R01MH070741 (NIH)
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Complicated Grief
Keywords: Grief; Bereavement; Psychotherapy; Randomized controlled trial; Treatment study

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complicated Grief Treatment (Experimental): Targeted psychotherapy for complicated grief
  Interventions: Behavioral: Complicated Grief Treatment
- Interpersonal Therapy (Active Comparator): Standard IPT is a comparator treatment
  Interventions: Behavioral: Interpersonal Therapy

INTERVENTIONS:
Behavioral: Complicated Grief Treatment — Complicated Grief Treatment (CGT) is a targeted psychotherapy for complicated grief. The treatment integrates principles, strategies and techniques from interpersonal psychotherapy, trauma-focused cognitive behavioral treatment and motivational interviewing. Treatment includes 16 sessions provided weekly.
  Other Names: CGT
  Arms: Complicated Grief Treatment
Behavioral: Interpersonal Therapy — Standard form of interpersonal psychotherapy delivered for 16 sessions weekly.
  Other Names: IPT
  Arms: Interpersonal Therapy

SUMMARY:
A comparison study of 16 week treatment with either specialized psychotherapy for complicated grief (CGT) or with standard interpersonal psychotherapy (IPT) in older adults with complicated grief.

DETAILED DESCRIPTION:
According to the National Council on Aging (1), in 2005, there were more than 10 million older Americans who were widowed (8.6 million women (43%) and 2.1 million men (14%) over the age of 65). These people are at risk for a debilitating reaction called Traumatic or Complicated Grief (CG: the term now used for this condition). Studies confirm that Complicated Grief can be reliably identified and occurs in about 10-20% of bereaved individuals. CG appears to carry much of the risk for negative outcomes of bereavement. CG can affect health status and influence decisions about personal health care. The risk of hypertension is 10 times greater among widowed subjects who meet consensus criteria for CG compared to those who do not, while subjects with CG are 17 times less likely to have visited a physician in the months since the death. Despite its high prevalence and significant morbidity, there are no proven efficacious treatments. The PI of this project developed a novel psychotherapy called Complicated Grief Treatment (CGT), and has now completed a study (MH60783) comprised of adults over age 18, that confirmed efficacy of this approach. Participants ≥ age 60 (n=29) were less likely to be employed and more likely to live alone. We observed better response to CGT than IPT, as in younger adults. However, confirmation of efficacy among seniors is important, since older people have different vulnerabilities and different problems in adjusting to grief than younger adults. We plan to conduct a randomized controlled study of CGT v IPT in individuals > 50 years of age who meet criteria for complicated grief and have no contraindications to study participation. Our specific aims are: 1) To compare results of 16 sessions of either CGT or standard IPT. We hypothesize that CGT will produce a higher response rate and shorter time to response than IPT, and that responders will show significantly greater reduction in associated symptoms and impairment than non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Complicated Grief is the most important problem
* Ability to give informed consent
* Fluent in English
* Willingness to have sessions audiotaped
* Willing to undergo random assignment

Exclusion Criteria:

* Diagnosis of one or more of the following disorders: Schizophrenia or other psychotic disorder, current (past 6 months) substance abuse or positive urine toxicology exam, Bipolar Disorder, current manic episode, Dementia
* Acute, unstable or severe medical illness such as (but not limited to) stroke, epilepsy, or other neurodegenerative disorders, metastatic or active cancer, hepatic disease, or primary renal disease requiring dialysis
* Pending or active disability claim or lawsuit related to the death
* Concurrent psychosocial therapy
* Judged to be at serious risk to self or others
* For people currently taking antidepressant medications, to be included in the study they must be on the medication for at least 3 months and for at least 6 weeks on the same dose

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2008-03; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Responder status on Complicated Grief Clinical Global Impression-Improvement (CGI-I) Scale | Week 20
  Brief rating scale frequently used in clinical trials. For this study, version modified for complicated grief will be used. The rating will be done by the Independent Evaluator.

SECONDARY OUTCOMES:
Change in score on Inventory of Complicated Grief (ICG) Scale | Up to 48 weeks from baseline
  The ICG is a 19-item self-report instrument that assesses symptoms of CG. This scale has been utilized previously in treatment studies of CG. Random regression model will be applied to evaluate the score trajectory from baseline to week 20 and from week 20 to week 48.
Change in score on Work and Social Adjustment Scale (WSAS) | Up to 48 weeks from baseline
  The WSAS is a modification of a scale introduced by Hafner and Marks (1976), consisting of 0-8 point ratings of the extent to which symptoms interfere with five areas of daily functioning: work, home management, private leisure, social leisure, and family relationships. It is a well-validated, widely used self-report measure. Random regression model will be applied to evaluate the score trajectory from baseline to week 20 and from week 20 to week 48.
Change in score on Grief Related Avoidance Questionnaire (GRAQ) Scale | Up to 48 weeks from baseline
  GRAQ is a questionnaire developed by the study investigators to elicit information related to avoidance of common situations and activities following the death. This scale has good psychometric properties and will be used to assess avoidance as a possible moderator predicting better outcome with CGT. It will be analyzed using random regression model.
Change in results from Structured Interview for Complicated Grief (SCI-CG) | Up to 16 weeks from baseline
  The SCI-CG is a clinician-administered structured interview developed for the study. It includes a composite of diagnostic criteria proposed by Horowitz and Prigerson. The interview was piloted and refined in the initial phase of current study.
Change in results on Typical Beliefs Questionnaire (TBQ) | Up to 16 weeks from baseline
  TBQ is a 34 item questionnaire evaluating how strongly subjects endorse certain beliefs that are common during bereavement related to self, the relationship, and perceptions of the world.

CONTACTS AND LOCATIONS:
Overall Officials: M. Katherine Shear, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Shear K, Frank E, Houck PR, Reynolds CF 3rd. Treatment of complicated grief: a randomized controlled trial. JAMA. 2005 Jun 1;293(21):2601-8. doi: 10.1001/jama.293.21.2601. PMID 15928281
- [Derived] Lechner-Meichsner F, Mauro C, Skritskaya NA, Shear MK. Change in avoidance and negative grief-related cognitions mediates treatment outcome in older adults with prolonged grief disorder. Psychother Res. 2022 Jan;32(1):91-103. doi: 10.1080/10503307.2021.1909769. Epub 2021 Apr 5. PMID 33818302
- [Derived] Ghesquiere A, Theresa Schwartz, Wang Y, Mauro C, Skritskaya N, Shear MK. Performance and psychometric properties of the Interpersonal Support Evaluation List (ISEL) in older adults with Complicated Grief. J Affect Disord. 2017 Aug 15;218:388-393. doi: 10.1016/j.jad.2017.05.004. Epub 2017 May 7. PMID 28501738
- [Derived] Shear MK, Wang Y, Skritskaya N, Duan N, Mauro C, Ghesquiere A. Treatment of complicated grief in elderly persons: a randomized clinical trial. JAMA Psychiatry. 2014 Nov;71(11):1287-95. doi: 10.1001/jamapsychiatry.2014.1242. PMID 25250737
- See also: Study website — http://www.complicatedgrief.org/